CLINICAL TRIAL: NCT04238052
Title: Evaluation of the Ability of Non-invasive Blood Pressure Measurement in the Dependent and Non-dependent Upper Extremities for Detecting Intra-operative Hypotension in the Lateral Position
Brief Title: Assessing the Ability of Non-invasive Blood Pressure Measurement in Both Arm for Detecting Hypotension in the Lateral Position
Status: Completed | Type: Observational
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Maha Mostafa Ahmad, MD, Principal Investigator, Kasr El Aini Hospital
Other Study IDs: MS-257-2019
Record Dates: First submitted 2020-01-19; First posted 2020-01-23 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Non-invasive Blood Pressure; Hypotension
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Intra-operative hypotension is linked to increased postoperative morbidity and mortality. Intra-operative MAP below 60-70 mmHg or SBP below 100 mmHg increase the risk of post operative myocardial injury, acute kidney injury and death. accurate measurement of blood pressure is fundamental in proper mangement of intraperative hypotension.

Measurement of arterial blood pressure through an arterial catheter is restricted to patients with major, rapid changes in blood pressure in the operating room as well as the intensive care units. Among non-invasive blood pressure (NIBP) monitors, oscillometric blood pressure measuring technology is considered the standard and the most widely used method in medical practice. In oscillometric blood pressure monitor, a pressure transducer located in the cuff senses the maximal arterial oscillation, which represents the mean arterial pressure, and according to the device's algorithm the systolic and diastolic blood pressure (SBP and DBP) will be calculated.

The upper arm is the standard location of application of the blood pressure cuff as it is aligned with the heart level regardless the patient position. Many surgical procedures, sometimes major, are conducted in the lateral position; during these operations, the choice of the side for application of the NIBP cuff is a challenging decision with no clear recommendations. The non-dependent upper limb is claimed to be inaccurate measurement site because the cuff position is above the level of the heart. While, the dependent upper limb might be affected by compression of the axilla and the upper arm. No data, to the best of our knowledge are available for the accuracy of NIBP in both upper limbs in the lateral position using the invasive arterial blood pressure (IBP) as a reference for detecting intraoperative hypotension.

DETAILED DESCRIPTION:
Preoperatively, the upper limb circumference will be measured at the mid arm, and the NIBP cuff size will be selected according to the recommendations of American Heart Association (cuff length and width will be 80% and 40% of arm circumference respectively) Upon arrival to the operating room, a non-invasive blood pressure (NIBP) reading will be obtained in both upper limbs in supine position. Patients with difference of 10 mmHg or above between both limbs will be excluded from the study.

Induction of general anesthesia will be achieved by administration of 2 mg/kg propofol, 2 mcg/kg fentanyl and 0.5 mg/kg atracurium. A 20 G radial arterial catheter will be inserted in the upper limb which is planned to be dependent. The arterial catheter will be connected to a pressure transducer at the level of the heart. Supine IBP reading will be recorded 5-minutes after intubation of the trachea in the supine position with simultaneous NIBP in both upper limbs at 3-minutes intervals. Five-minutes after settling in the lateral position, NIBP will be obtained alternating between the dependent and non-dependent limbs at 5-minutes intervals till the end of the operation or till reaching a maximum of 10 readings from each side.

The reading of the IBP will be obtained from the contralateral upper limb during inflation of the cuff of the NIBP. Whilst, the reading of the IBP will be obtained from the same upper limb just before the inflation of the cuff of the NIBP

ELIGIBILITY:
Inclusion Criteria:

* adult patients (18-60 years)
* American Society of Anesthesiologist - Physical Status I-II,
* scheduled for elective non-cardiac surgery under general anesthesia and invasive blood pressure monitoring is part of their intraoperative management

Exclusion Criteria:

Patients with any of the following morbidities:

* peripheral vascular diseases,
* upper limb operations,
* upper limb scars,
* upper limb deep venous thrombosis, and
* arrhythmias

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: adult patients (18-60 years), American Society of Anesthesiologist - Physical Status I-II, scheduled for elective non-cardiac surgery under general anesthesia and invasive blood pressure monitoring is part of their intraoperative management
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2020-01-23 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
accuracy of MAP measurement at dependent arm for detectiong intraoperative hypotension at lateral position | up to 100 minutes
  MAP below 70 mmHg

SECONDARY OUTCOMES:
accuracy of MAP measurement at non-dependent arm for detectiong intraoperative hypotension at lateral position | 5 minutes after settling in the lateral position, every 5 minutes for 100 minutes
  MAP below 70 mmHg
accuracy of SBP measurement at dependent arm for detectiong intraoperative hypotension at lateral position | 5 minutes after settling in the lateral position, every 5 minutes for 100 minutes
  SBP below 100 mmHg
accuracy of SBP measurement at non-dependent arm for detecting intraoperative at lateral position | 5 minutes after settling in the lateral position, every 5 minutes for 100 minutes
  SBP below 100 mmHg
correlation between NIBP measurement at dependent arm in relation to invasive blood at lateral position pressure | 5 minutes after settling in the lateral position, every 5 minutes for 100 minutes
  mmHg
mean bias and agreement between NIBP measurement at dependent arm in relation to invasive blood at lateral position pressure | 5 minutes after settling in the lateral position, every 5 minutes for 100 minutes
  mmHg
correlation between NIBP measurement at non-dependent arm in relation to invasive blood at lateral position pressure | 5 minutes after settling in the lateral position, every 5 minutes for 100 minutes
  mmHg
mean bias and agreement between NIBP measurement at non-dependent arm in relation to invasive blood at lateral position pressure | 5 minutes after settling in the lateral position, every 5 minutes for 100 minutes
  mmHg

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alaini Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mostafa M, Hasanin AM, Elsayed OS, Mostafa MM, Sarhan K. Accuracy of oscillometric blood pressure measurement at both arms in the lateral position. Blood Press Monit. 2021 Oct 1;26(5):364-372. doi: 10.1097/MBP.0000000000000546. PMID 34001758